CLINICAL TRIAL: NCT05410951
Title: LobularCard Trial: Searching for Novel Germline Mutations in Lobular Breast Cancer Patients
Acronym: LobularCard
Status: Active, not recruiting | Type: Observational
Sponsor: European Institute of Oncology (Other)
Responsible Party: Sponsor
Other Study IDs: IEO 1730
Record Dates: First submitted 2022-06-06; First posted 2022-06-08 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Lobular Breast Carcinoma; Lobular in Situ Breast Carcinoma; BRCA1 Mutation; BRCA2 Mutation
MeSH Terms: conditions — Carcinoma, Lobular; Breast Carcinoma In Situ

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The screening analysis will be performed on blood samples available in European Institute of Oncology Biobank by Next Generation Sequencing (NGS) technology using the TruSight Hereditary Cancer panel (Illumina) to analyze the entire coding regions of 113 genes selected genes and 125 SNPs, starting from 50 ng of gDNA extracted with MagCore HF16 Plus (Diatech Labline).
  Libraries will be constructed following the manufacturer protocols (Nextera Flex for Enrichment Illumina) and will be sequenced with Illumina MiSeq Sequencer or Illumina NextSeq Sequencer available in the laboratory.
  Data will be analyzed with a dedicated software. Finally, all mutations will be confirmed using the Sanger sequencing method (3500xL Dx Genetic Analyzer, Thermo Fisher Scientific).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Illumina panel — Determination of germline mutations using a recent panel including 113 genes from the "Illumina" protocol

SUMMARY:
This is a cross-sectional and retrospective study of a cohort of patients with invasive lobular breast cancer (LBC) or in situ lobular neoplasia (LIN3).

The main endpoint is the relative frequency of patients with a germline mutation using a recent panel including 113 genes from the "Illumina" protocol.

In case of identification of a novel pathogenetic germline mutations, a personalized follow-up will be offered to each patient (in case of genes at moderate-, low-penetrance), or prophylactic mastectomy (in case of genes at high-penetrance).

Breast screening in moderate-, low-penetrance mutated patients should be performed periodically using digital mammography, ultrasound and MRI, and will be routinely observed.

Patients will be scheduled for follow-up at six-month intervals for 5 years at our outpatient clinic, and yearly thereafter

DETAILED DESCRIPTION:
Pathogenic or likely pathogenic variants (commonly referred to as mutations) in high-penetrance breast cancer (BC) susceptibility genes increase the risk of BC more than fourfold. Germline mutations in BRCA1 or BRCA2 (BRCA1/2) are found in 3% to 4% of all women with BC, including 10% to 20% of those with triple-negative breast cancer (TNBC) and 10% to 15% of Jewish women with BC.

Recent international guidelines consider only a small group of gene as high-penetrance risk: BRCA1/2, CDH1, PTEN, and PALB2 [2], the remaining are classified as moderate-, low-penetrance risks.

There are no specific associations between these germline mutations and BC histotypes. In accord with recent genetic results reported in literature, lobular histotype seems associated with a specific germline pathway.

We hypothesize that other genes are associated with a susceptibility for lobular breast carcinoma (LBC) predisposition and that novel genetic factors should be described, especially in subjects with early onset of LBC.

In this context we selected a recent panel including 113 genes from the "Illumina" protocol.

The screening analysis will be performed by Next Generation Sequencing (NGS) technology using the TruSight Hereditary Cancer panel (Illumina) to analyze the entire coding regions of 113 genes selected genes and 125 SNPs, starting from 50 ng of gDNA extracted with MagCore HF16 Plus (Diatech Labline).

The proposed project is scheduled in three major tasks:

1) Data collection, including family history assessment and pedigree analysis for eligible subjects deserving genetic screening; 2) Genomic characterization of LBC in subjects with germline mutation; 3) Evaluation of disease-free survival and overall survival in subjects with germline mutation and establishment of a specific clinical follow-up for these patients.

ELIGIBILITY:
Inclusion criteria:

1. All LBC observed retrospectively at the European Institute of Oncology, with a proved diagnosis of LBC (biopsy or operated)
2. Patients with blood available in biobank Exclusion criteria

   * Patients with a previous cancer (except skin basal cell carcinoma)
   * Patients with ductal or mixed BC

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with in situ (LIN3) or invasive LBC or bilateral LBC or LBC with or without family history for BC, with blood sample available in European Institute of Oncology biobank
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2022-05-16 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-05-16 (Estimated)

PRIMARY OUTCOMES:
Relative frequency of patients with a germline mutation | 1 month
  Frequency of germline mutation status in patients with in situ (LIN3) or invasive LBC or bilateral LBC or LBC with or without family history for breast cancer

SECONDARY OUTCOMES:
Correlation of clinic-pathological data between genes at high-penetrance versus other genes | 1 month
  correlation of clinic-pathological data between genes at high-penetrance (BRCA1/2, CDH1, PTEN, and PALB2) vs. other genes
Prevalence of germline mutation status by clinical strata | 1 month
  Prevalence of germline mutation status by early onset LBC (age <45 years), bilateral LBC, LBC with family history for breast cancer
Association with disease free survival and overall survival | 5 years
  prognostic role of mutation status: the association with disease free survival and overall survival
Association of mutation status with molecular subtypes | 3 months
  association of mutation status with molecular subtype of primary tumor (Luminal A, Luminal B, Basal-like, HER2-enriched)

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Corso, PhD, MD, Principal Investigator — European Institute of Oncology
Locations (1):
- European Institute of Oncology, Milan, Italy

IPD SHARING:
Plan to Share IPD: No